CLINICAL TRIAL: NCT02666378
Title: Imaging Markers of Subclinical Cardiotoxicity in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Heart Association (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Reza Nezafat, Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 15-017
Record Dates: First submitted 2015-11-16; First posted 2016-01-28 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CMR/ECHO: Prior to starting chemotherapy treatment, the participant will undergo the following procedures:
  * Cardiac Magnetic Resonance Imaging (CMR)
  * Echocardiogram (ECHO) in patients with no clinically indicated scans
  * Each imaging procedure will be repeated at predetermined times during the protocol
  * Simple blood collection for plasma biomarker analysis
  Interventions: Other: Cardiac Magnetic Resonance Imaging (CMR); Other: Echocardiogram (ECHO)

INTERVENTIONS:
Other: Cardiac Magnetic Resonance Imaging (CMR) — Subjects will be recruited for observational cardiac magnetic resonance imaging.
  Other Names: MRI
Other: Echocardiogram (ECHO) — Subjects will undergo a research echocardiogram if a clinical echocardiogram has not already been ordered.

SUMMARY:
This research study is evaluating the use of Cardiac Magnetic Resonance Imaging (CMR) as a method of detecting early signs of damage to the heart that can be associated with anthracycline-based chemotherapy for the treatment of breast cancer.

DETAILED DESCRIPTION:
One of the side effects observed in breast cancer patients receiving anthracycline-based treatment is heart complications in which the heart muscle is weakened and no longer able to pump sufficient amounts of blood throughout the body. This complication can lead to the following symptoms: shortness of breath on exertion, swollen ankles and feet, lack of energy and a reduced capacity to carry out day-to-day activities.

This research study is focused on identifying the early signs of such heart complications using CMR, which may allow preventative treatment options to be made available in future.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Have histologic diagnosis of breast carcinoma
* Scheduled to receive standard clinical therapy designed by their treating oncologist
* Patients should receive anthracycline as part of the recommended treatment
* Able to give informed consent.

Exclusion Criteria:

* Contraindication to contrast CMR including eGFR <30 mls/min/1.73m2
* Uncontrolled serious concurrent illness
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Cardiotoxicity | 1 year after completion of treatment
  Cardiotoxicity as measured by changes in left ventricular ejection fraction within one-year of completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Reza Nezafat, Ph.D, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States